CLINICAL TRIAL: NCT02414451
Title: Trial of Propranolol in Adults and Adolescents With Autism Spectrum Disorder (ASD) and Predictors of Response
Brief Title: Trial of Propranolol in Adults and Adolescents With ASD and Predictors of Response
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No need for a pilot study. New study will be opened.
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, David Beversdorf, Associate Professor, Radiology, Neurology, and Psychology, University of Missouri-Columbia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 200089
Record Dates: First submitted 2015-03-20; First posted 2015-04-10 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Autism
Keywords: Propranolol
MeSH Terms: conditions — Autistic Disorder | interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propranolol arm (Experimental): Propranolol will be administered via oral capsule(s) daily for a period of 10 weeks, involving gradual titration up from 40mg to 100mg and subsequent tapering off of the drug. The titration/tapering schedule will be as follows:
  Week 1: 40 mg propranolol (1 capsule, nightly) Week 2: 80 mg propranolol (2 40mg capsules, morning & night) Weeks 3 - 8: 100 mg propranolol (3 capsules, 40 mg/morning, 20mg/afternoon, & 40mg/night) Week 9: 60 mg propranolol (2 capsules, 40 mg/morning & 20mg/night) Week 10: 20 mg propranolol (1 capsule, nightly) Week 11: no capsules
  Interventions: Drug: Propranolol
- Placebo arm (Placebo Comparator): Placebo will be administered via lactose-filled oral capsule(s) daily for a period of 10 weeks. The schedule of placebo administration will be as follows:
  Week 1: 1 capsule, nightly Week 2: 2 capsules, morning & night Weeks 3 - 8: 3 capsules, morning, afternoon, & night Week 9: 2 capsules, morning & night Week 10: 1 capsule, nightly Week 11: no capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propranolol — Week 1: 40 mg propranolol (1 capsule, nightly) Week 2: 80 mg propranolol (2 40mg capsules, morning & night) Weeks 3 - 8: 100 mg propranolol (3 capsules, 40 mg/morning, 20mg/afternoon, & 40mg/night) Week 9: 60 mg propranolol (2 capsules, 40 mg/morning & 20mg/night) Week 10: 20 mg propranolol (1 capsule, nightly) Week 11: no capsules
  Other Names: Inderal
  Arms: Propranolol arm
Drug: Placebo — Placebo will be administered via lactose-filled oral capsule(s) daily for a period of 10 weeks. The schedule of placebo administration will be as follows:
  Week 1: 1 capsule, nightly Week 2: 2 capsules, morning & night Weeks 3 - 8: 3 capsules, morning, afternoon, & night Week 9: 2 capsules, morning & night Week 10: 1 capsule, nightly Week 11: no capsules
  Arms: Placebo arm

SUMMARY:
The purpose of this study is to explore the effects of propranolol on social interaction, and secondarily on language, anxiety, adaptive behaviors, and global function in high functioning adults and adolescents with autism in a double-blinded, placebo-controlled pilot trial.

DETAILED DESCRIPTION:
The investigators' specific aim is to examine the effects of serial doses of propranolol on social interaction, and secondarily on language tasks, anxiety, adaptive behaviors, and global function in high functioning adults and adolescents with autism in a double-blinded, placebo-controlled trial. The investigators will also examine whether response to treatment can be predicted based upon markers of autonomic functioning, such as skin conductance and heart rate variability, and whether anxiety predicts treatment response. The investigators' hypothesis is that social functioning and language abilities will benefit from serial doses of propranolol, as the investigators have demonstrated in previous single-dose studies. The investigators also predict that those with the greatest degree of autonomic dysregulation will demonstrate the greatest benefit from the drug.

ELIGIBILITY:
Inclusion Criteria:

* For participants with autism: High-functioning, native-English speaking subjects with ASD aged 15-30. High-functioning ASD is defined in this study by the DSM-V criteria plus Autism Diagnostic Interview-Revised (ADI-R) criteria for Autism, and Wechsler Abbreviated Scales of Intelligence (WASI) full scale IQ of at least 85.

Exclusion Criteria:

* For participants with autism: Non-autism learning disability (e.g. dyslexia),
* major psychiatric diagnosis (e.g. major depression, schizophrenia, bipolar disorder),
* other neurological diagnosis,
* major head trauma,
* any of the following exclusionary criteria related to propranolol (diabetes, reactive airway/pulmonary disease, thyroid disease, bradyarrhythmias, unexplained syncope, narrow angle glaucoma, pregnancy, known hypersensitivity/adverse reaction to beta-blockers),
* any of the following exclusionary criteria related to placebo (severe allergy to lactose),
* any of the following exclusionary criteria related to the psychophysiological measurements (history of rash from adhesives).

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in General Social Outcome Measure (GSOM) | Week 1, Week 4, Week 8, Week 12, Week 15, Week 19
  The GSOM is a brief evaluation tool that measures a participant's level of social functioning and how it changes with intervention. There GSOM includes 4 different tasks: conversational reciprocity, ability to recognize facial expressions, social problem solving, affect demonstration, and emotional perspective taking. The experimenter administers each component of the GSOM to the participant and then scores their responses according to a pre-determined scoring rubric. Each component is scored on a 1-5 or 0 - 2 scale, with higher total scores indicating better social functioning. A video camera will be used to record the participant's behavior during GSOM administration for the purposes of having two independent raters score the tasks after the study session is complete. The video camera will be turned off for the remainder of the study session. A camera will also be used during the affect demonstration task of the GSOM.
Change in Social Responsiveness Scale (SRS) | Week 1, Week 4, Week 8, Week 12, Week 15, Week 19
  This 65-item, parent-report measure asks questions about a participants' social awareness, social information processing, capacity for reciprocal social responses, social anxiety or avoidance, and characteristic autistic preoccupations or traits.

SECONDARY OUTCOMES:
Change in Anagrams task | Week 1, Week 4, Week 8, Week 12, Week 15, Week 19
  To assess verbal problem solving, participants will be given a set of 20 anagram s (scrambled words, where letters are rearranged to form a word: e.g., IRCKB → BRICK). A maximum of 120 seconds will be allowed for each anagram. Number solved and solution latency (with failed anagrams recorded as 120 seconds) will be recorded.
Change in Verbal fluency for categories task | Week 1, Week 4, Week 8, Week 12, Week 15, Week 19
  To assess verbal and semantic fluency, participants will be asked to generate as many words as possible within one minute each from three different categories (e.g. animals, things to wear, vegetables). Total number of distinct words (not including proper nouns) will be recorded for each session.
Change in Spence Children's Anxiety Scale (SCAS) | Week 1, Week 4, Week 8, Week 12, Week 15, Week 19
  To assess anxiety, the SCAS will be completed by the participants. This self-report measure yields a total score in addition to six subscales (separation anxiety, social phobia, obsessive compulsive, panic/agoraphobia, physical injury fears, and generalized anxiety).
Vertical attention task | Week 1
  At the initial study visit only, a vertical spatial attention task will be administered to assess whether individuals with ASD display a vertical attention bias. A 4'x 3' board will be hung in the exam room in the landscape orientation, and the experimenter will present a total of 72 lines on the board for the participant to bisect or quadrisect (i.e., "place a mark in the middle of the line" or "place a mark that is one quarter or 25% from the top or bottom of the line") with a pen at one of three spatial positions (above eye level, eye level, below eye level).
Change in Clinical Global Impression of Change (CGIC) scale | Week 4, Week 8, Week 12, Week 15, Week 19
  To assess overall changes in the participant's ASD-related clinical symptoms, the CGIC will be administered. The CGIC consists of a 7-point subjective scale assessing change from baseline. On this scale, scores of 1, 2, and 3 represent marked, moderate, and mild improvement, respectively. A score of 4 represents no change. Scores of 5, 6, and 7 represent mild, moderate, and marked worsening, respectively. CGIC scores from both the parent/caregiver and the blinded PI (licensed physician) will be utilized.
Change in Autism Impact Measure (AIM) | Week 1, Week 4, Week 8, Week 12, Week 15, Week 19
  The AIM will be administered to assess the frequency and impact of a participant's ASD-related symptoms. A parent/caregiver is asked a series of 41 questions regarding the frequency and the impact, or interference resulting from, a series of autism-associated behaviors. Overall impact and frequency scores, as well as subscale scores, will be obtained from this measure.
Change in Vineland Adaptive Behavior Scales-II (VABS) | Week 1, Week 4, Week 8, Week 12, Week 15, Week 19
  To assess overall adaptive functioning, the VABS will be administered in the form of a structured interview with the parent/caregiver. The VABS is a well validated assessment used for the full range of our subjects' ages and yields standard scores in Communication, Daily Living Skills, Socialization, and Motor Skills. VABS scores for Communication, Daily Living Skills, and Socialization will be monitored in this study.
Change in Aberrant Behavior Checklist (ABC) | Week 1, Week 4, Week 8, Week 12, Week 15, Week 19
  To assess overall behavioral disturbances, a parent/caregiver of the participants will complete ABC. This 58-item questionnaire is a well validated, reliable, and widely used assessment tool for interventions for a range of cognitive disorders.
Change in Clinical Global Impression of Severity (CGIS) scale | Week 1, Week 4, Week 8, Week 12, Week 15, Week 19
  To assess overall severity of a participant's ASD-related clinical symptoms, the CGIS will be administered. The CGIS consists of a 7-point subjective scale assessing symptom severity. On this scale, scores of 1, 2, and 3 represent normal, some presence of symptoms, and mild behavior, respectively. A score of 4 represents moderate behavior. Scores of 5, 6, and 7 represent marked, severe, and among the most severe behavior, respectively. CGIS scores from both the parent/caregiver and the blinded PI (licensed physician) will be utilized.

CONTACTS AND LOCATIONS:
Overall Officials: David Q Beversdorf, MD, Principal Investigator — University of Missouri-Columbia